CLINICAL TRIAL: NCT00162396
Title: Evaluation of Genetic Factors That May Account for Variability in the Response to Salbutamol Among Patients Suffering From Asthma
Brief Title: Genetic Determinants of the Response to Salbutamol Among Asthma Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hadassah Medical Organization (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: yc195511-HMO-CTIL
Record Dates: First submitted 2005-09-11; First posted 2005-09-13 (Estimated); Last update posted 2008-10-29 (Estimated); Status verified 2008-10

CONDITIONS: Asthma
Keywords: Albuterol; β2 Adrenergic receptor; Polymorphism
MeSH Terms: conditions — Asthma | interventions — Albuterol

INTERVENTIONS:
Drug: Albuterol

SUMMARY:
The response to salbutamol varies greatly among individuals. Data from previous studies indicate that some of the variability is accounted for by genetic polymorphisms in the gene encoding for the adrenoceptor subtype β2. The current study was designed to evaluate variability in the response to salbutamol among recently diagnosed patients who have not been treated by β2 agonists or corticosteroids.

Lung function tests will be performed prior to and following a single dose administration of salbutamol through inhalation. Additional pharmacodynamic indices will be monitored including pulse and blood pressure. Three samples of plasma will be drawn for the evaluation of salbutamol plasma concentration.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Recently diagnosed as asthmatic

Exclusion Criteria:

* Current treatment by β2 agonist
* Current treatment by corticosteroids
* Acute asthma attack

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 1999-08

PRIMARY OUTCOMES:
Change in lung function tests after salbutamol inhalation
Change in blood pressure and pulse after salbutamol inhalation

CONTACTS AND LOCATIONS:
Overall Officials: Yoseph Caraco, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel